CLINICAL TRIAL: NCT05881252
Title: An Observational Study of Perinatal Outcomes Following Change in Clinical Criteria in for Treatment of Maternal Hypertension
Brief Title: Perinatal Outcomes Following Change in Clinical Criteria in for Treatment of Maternal Hypertension
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kristen Cagino, Fellow, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-23-0241
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Maternal Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional clinical blood pressure threshold of SBP >= 160 mmHg for acute treatment of hypertension
  Interventions: Procedure: Clinical blood pressure threshold of SBP >= 160 mmHg for acute treatment of hypertension
- Updated clinical blood pressure threshold of SBP >= 180 mmHg for acute treatment of hypertension
  Interventions: Procedure: Clinical blood pressure threshold of SBP >= 180 mmHg for acute treatment of hypertension

INTERVENTIONS:
Procedure: Clinical blood pressure threshold of SBP >= 160 mmHg for acute treatment of hypertension — Patients are treated for hypertension if SBP >= 160 mmHg.
  Groups: Traditional clinical blood pressure threshold of SBP >= 160 mmHg for acute treatment of hypertension
Procedure: Clinical blood pressure threshold of SBP >= 180 mmHg for acute treatment of hypertension — Patients are treated for hypertension if SBP >= 180 mmHg.
  Groups: Updated clinical blood pressure threshold of SBP >= 180 mmHg for acute treatment of hypertension

SUMMARY:
The purpose of this study is observe outcomes before and after a change in clinical practice in the threshold for management of severe hypertension in pregnancy and the post-partum period. Outcomes will be observed for 10 months under the current (traditional) clinical blood pressure threshold for acute treatment of hypertension, which is >= 160 millimeters of mercury (mmHg) systolic blood pressure (SBP). This will be followed by one month of education about rationale for the new SBP threshold of >= 180 mmHg and change of clinical guidelines. Then, there will be 10 months of observation after adopting the updated clinical threshold for acute antihypertensive treatment (>= 180 SBP).

ELIGIBILITY:
Inclusion Criteria:

* any individual > 20 weeks' gestation in triage or admitted at Children's Memorial Hermann Hospital (CMHH) and with blood pressure with >= 160/110 mmHg

Exclusion Criteria:

* Active seizure, stroke, Congestive Heart Failure (CHF)/pulmonary edema, acute kidney injury (AKI), or myocardial infarction (MI)
* A history of stroke, CHF, chronic kidney disease (CKD), MI
* Have Hemolysis, elevated liver enzymes, low platelets (HELLP) syndrome or thrombocytopenia (platelets < 100×10^9/L)
* Persistent neurologic symptoms including headache >8/10 one hour after analgesic or blurry vision/loss of vision

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual > 20 weeks' gestation in triage or admitted at Children's Memorial Hermann Hospital (CMHH) in Houston, Texas and with blood pressure with >= 160/110 mmHg
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with Congestive Heart Failure/Pulmonary Edema, hemorrhagic or ischemic Stroke, Acute Kidney Injury (creatinine > 1.5mg/dL), and/or or Myocardial Ischemia. | during the time of delivery hospitalization (about 2 days to 3 months)
  The primary outcome is a composite outcome, and will be reported as number of patients who have Congestive Heart Failure/Pulmonary Edema, hemorrhagic or ischemic Stroke, Acute Kidney Injury (creatinine > 1.5mg/dL), and/or Myocardial Ischemia.

SECONDARY OUTCOMES:
Number of patients with non-reassuring fetal heart rate tracing (NR-FHRT) requiring caesarean delivery | at the time of delivery
Number of patients with Apgar score < 7 at 5 min | 5 minutes after birth
  The Apgar score indicates the status of the newborn infant immediately after birth. Apgar score ranges from 0-10, with a higher score indicating a better outcome.
Number of patients with eclampsia | during the time of delivery hospitalization (about 2 days to 3 months)
Number of patients with placental abruption | during the time of delivery hospitalization (about 2 days to 3 months)
Number of patients with posterior reversible encephalopathy syndrome (PRES) | during the time of delivery hospitalization (about 2 days to 3 months)
Number of patients with hemolysis, elevated liver enzymes, low platelets (HELLP) syndrome | during the time of delivery hospitalization (about 2 days to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Cagino, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UT Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No